CLINICAL TRIAL: NCT04946721
Title: 2177GCCC: Identifying Novel Treatment Targets and Biomarkers for Ocular Surface Disease in Patients With Ocular Graft vs Host Disease (oGVHD) a Biobank Study
Brief Title: 2177GCCC:ID'Ing tx Targets and Biomarkers for Ocular Surface Disease in Pt w/ oGVHD
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Other Study IDs: 2177GCCC
Record Dates: First submitted 2021-06-15; First posted 2021-07-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease; oGVHD
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Certain biological specimens (ocular surface wash, mucocellular material, corneal filaments or impression cytology, or blood) will be collected and stored and analyzed to obtain immunologic, cellular, or molecular mechanistic insights into the patient's disease processes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1.BMT Patients (Study): Patients prior to receiving a bone marrow transplant will be recruited during their initial intake prior to their BM transplant through the PI's regularly scheduled appointment with these patients.
  Interventions: Diagnostic Test: The standard care exam and biological specimens' collection
- 2.Controls: Patients with no history of eye disease or cancer history
  Interventions: Diagnostic Test: The standard care exam and biological specimens' collection

INTERVENTIONS:
Diagnostic Test: The standard care exam and biological specimens' collection — During each visit, in addition to standard of care exams, certain biological specimens ( ocular surface wash, mucocellular material, corneal filaments or impression cytology of conjunctiva, blood or serum) will be collected.

SUMMARY:
Evaluate and study the immunologic changes to the ocular surface in cancer patients.

DETAILED DESCRIPTION:
This is a longitudinal natural history study to evaluate and study the immunologic changes to the ocular surface in cancer patients.

Two groups of subjects will be recruited for the study: 1) Pre-bone marrow transplant cancer patients. They will be evaluated every 3 months for 2 years.2) Normal control patients. They will be evaluated every 6 months for the duration of the study.

During each study visit, in addition to standard of care exams, certain biological specimens ( ocular surface wash, mucocellular material, corneal filaments, or impression cytology of conjunctiva, blood, or serum) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) who visit the Eye clinic either in the UMGCCC within the UMD Hospital or the UMD Faculty Physicians Ophthalmology Practice at the UMD Professional Building or satellite locations for initial visits or established visits.
* The patient must be able to understand and sign and date the informed consent form approved by the IRB.

Exclusion Criteria:

* Vulnerable populations: neonates, children, prisoners, institutionalized individuals.
* Inability or refusal to provide informed consent.
* History of ocular surgery (except refractive surgery or cataract surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of patients will be invited to participate in the study.
  1. BMT Patients (Study) - Patients prior to receiving a bone marrow transplant will be recruited during their initial intake prior to their BM transplant through the PI's regularly scheduled appointment with these patients.
  2. Controls - patients with no history of eye disease or cancer history.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Risk factors and markers for developing eye diseases | Up to 4 years
  Number of patients with the risks and markers who have developed the eye diseases during the study
2. The mechanisms of eye damage | Up to 4 years
  Number of patients who have eye damage during the study
The drug acting targets | Up to 4 years
  Number of patients who have eye diseases with eye surface changes after the treatment during the study.
The effect of ocular Graft-vs-Host Disease on the eye | Up to 4 years
  Number of patients who have eye surface changes with Graft-vs-Host Disease during the study

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sunshine, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Geenebaum Cancer Center, University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Sonawane S, Khanolkar V, Namavari A, Chaudhary S, Gandhi S, Tibrewal S, Jassim SH, Shaheen B, Hallak J, Horner JH, Newcomb M, Sarkar J, Jain S. Ocular surface extracellular DNA and nuclease activity imbalance: a new paradigm for inflammation in dry eye disease. Invest Ophthalmol Vis Sci. 2012 Dec 17;53(13):8253-63. doi: 10.1167/iovs.12-10430. PMID 23169882
- [Background] McDermott AM. New insight into dry eye inflammation. Invest Ophthalmol Vis Sci. 2012 Dec 17;53(13):8264. doi: 10.1167/iovs.12-11386. No abstract available. PMID 23248237
- [Background] Brinkmann V, Reichard U, Goosmann C, Fauler B, Uhlemann Y, Weiss DS, Weinrauch Y, Zychlinsky A. Neutrophil extracellular traps kill bacteria. Science. 2004 Mar 5;303(5663):1532-5. doi: 10.1126/science.1092385. PMID 15001782
- [Background] Cooper PR, Palmer LJ, Chapple IL. Neutrophil extracellular traps as a new paradigm in innate immunity: friend or foe? Periodontol 2000. 2013 Oct;63(1):165-97. doi: 10.1111/prd.12025. PMID 23931060
- [Background] Tibrewal S, Sarkar J, Jassim SH, Gandhi S, Sonawane S, Chaudhary S, Byun YS, Ivanir Y, Hallak J, Horner JH, Newcomb M, Jain S. Tear fluid extracellular DNA: diagnostic and therapeutic implications in dry eye disease. Invest Ophthalmol Vis Sci. 2013 Dec 11;54(13):8051-61. doi: 10.1167/iovs.13-12844. PMID 24255046
- [Background] Ogawa Y, Okamoto S, Wakui M, Watanabe R, Yamada M, Yoshino M, Ono M, Yang HY, Mashima Y, Oguchi Y, Ikeda Y, Tsubota K. Dry eye after haematopoietic stem cell transplantation. Br J Ophthalmol. 1999 Oct;83(10):1125-30. doi: 10.1136/bjo.83.10.1125. PMID 10502571
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Inamoto Y, Valdes-Sanz N, Ogawa Y, Alves M, Berchicci L, Galvin J, Greinix H, Hale GA, Horn B, Kelly D, Liu H, Rowley S, Schoemans H, Shah A, Lupo Stanghellini MT, Agrawal V, Ahmed I, Ali A, Bhatt N, Byrne M, Chhabra S, DeFilipp Z, Fahnehjelm K, Farhadfar N, Horn E, Lee C, Nathan S, Penack O, Prasad P, Rotz S, Rovo A, Yared J, Pavletic S, Basak GW, Battiwalla M, Duarte R, Savani BN, Flowers MED, Shaw BE, Petricek I. Ocular graft-versus-host disease after hematopoietic cell transplantation: Expert review from the Late Effects and Quality of Life Working Committee of the CIBMTR and Transplant Complications Working Party of the EBMT. Bone Marrow Transplant. 2019 May;54(5):662-673. doi: 10.1038/s41409-018-0340-0. Epub 2018 Dec 7. PMID 30531954
- [Background] Abud TB, Amparo F, Saboo US, Di Zazzo A, Dohlman TH, Ciolino JB, Hamrah P, Dana R. A Clinical Trial Comparing the Safety and Efficacy of Topical Tacrolimus versus Methylprednisolone in Ocular Graft-versus-Host Disease. Ophthalmology. 2016 Jul;123(7):1449-57. doi: 10.1016/j.ophtha.2016.02.044. Epub 2016 Apr 13. PMID 27086024
- [Background] An S, Raju I, Surenkhuu B, Kwon JE, Gulati S, Karaman M, Pradeep A, Sinha S, Mun C, Jain S. Neutrophil extracellular traps (NETs) contribute to pathological changes of ocular graft-vs.-host disease (oGVHD) dry eye: Implications for novel biomarkers and therapeutic strategies. Ocul Surf. 2019 Jul;17(3):589-614. doi: 10.1016/j.jtos.2019.03.010. Epub 2019 Apr 6. PMID 30965123
- [Background] Lelli GJ Jr, Musch DC, Gupta A, Farjo QA, Nairus TM, Mian SI. Ophthalmic cyclosporine use in ocular GVHD. Cornea. 2006 Jul;25(6):635-8. doi: 10.1097/01.ico.0000208818.47861.1d. PMID 17077652
- [Background] Kwon J, Surenkhuu B, Raju I, Atassi N, Mun J, Chen YF, Sarwar MA, Rosenblatt M, Pradeep A, An S, Dhall N, Mun C, Jain S. Pathological consequences of anti-citrullinated protein antibodies in tear fluid and therapeutic potential of pooled human immune globulin-eye drops in dry eye disease. Ocul Surf. 2020 Jan;18(1):80-97. doi: 10.1016/j.jtos.2019.10.004. Epub 2019 Oct 10. PMID 31606460